CLINICAL TRIAL: NCT06049992
Title: Stylet-driven vs. Lumenless Lead in Left-Bundle-Branch Pacing Randomized Trial
Brief Title: STylet-driven vs. LumenlEss Lead in Left-Bundle-Branch Pacing
Acronym: STYLE-LBBP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Puerta de Hierro University Hospital (Other)
Collaborators: Spanish Society of Cardiology (Other)
Responsible Party: Principal Investigator, Alvaro Lorente-Ros, Principal investigator, Puerta de Hierro University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STYLE-LBBP 2023
Record Dates: First submitted 2023-09-11; First posted 2023-09-22 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Left Bundle-Branch Pacing
Keywords: Left bundle-branch pacing; Conduction system pacing; Leadless; Stylet-driven pacing leads

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lumenless lead (Active Comparator): Left bundle branch stimulation using leads without internal lumen (Lumenless; Medtronic Selectsecure 3830, Minneapolis, USA).
  Interventions: Device: Pacemaker implantation with conduction system pacing using Lumenless leads
- Stylet-driven lead (Active Comparator): Left bundle branch pacing using leads with internal lumen and retractable helix (Tendril STS 2088TC, Abbott, Inc., USA; Solia S60, Biotronik, SE & Co., KG, Germany; Ingevity +, Boston Scientific, Marlborough, MA, USA).
  Interventions: Device: Pacemaker implantation with conduction system pacing using Stylet-driven leads

INTERVENTIONS:
Device: Pacemaker implantation with conduction system pacing using Lumenless leads — Pacemaker implantation for conduction system pacing will be done using leads without internal lumen (Lumenless; Medtronic Selectsecure 3830, Minneapolis, USA).
  Arms: Lumenless lead
Device: Pacemaker implantation with conduction system pacing using Stylet-driven leads — Pacemaker implantation for conduction system pacing will be done using leads with internal lumen and retractable helix (Tendril STS 2088TC, Abbott, Inc., USA; Solia S60, Biotronik, SE & Co., KG, Germany; Ingevity +, Boston Scientific, Marlborough, MA, USA)
  Arms: Stylet-driven lead

SUMMARY:
The STYLE-LBBP study aims to compare the efficacy and safety of left-bundle branch pacing between the two types of available pacing leads: lumenless vs stylet-driven.

DETAILED DESCRIPTION:
STYLE-LBBP is a randomized, non-blinded, multicenter clinical trial that compares the efficacy and safety of two types of available pacing leads in conduction system pacing (CSP). Patients referred to CSP who meet the inclusion and exclusion criteria will be enrolled and randomized into two groups: i)Left bundle branch pacing (LBBP) using leads without internal light (Lumenless; Medtronic Selectsecure 3830, Minneapolis, USA) or ii) LBBP with stylet-driven leads (Tendril STS 2088TC, Abbott, Inc., USA; Solia S60, Biotronik, SE & Co., KG, Germany; Ingevity +, Boston Scientific, Marlborough, MA, USA).

Efficacy in terms of achieving LBBP (selective and non-selective left bundle capture criteria) will be measured at implantation and after 24 hours. Complications of the procedure will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients referred for conduction system pacing

Exclusion Criteria:

* Patients with a prosthetic (metal or biologic) tricuspid valve.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2025-09-21 (Estimated); Study Completion 2025-09-22 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients in which left-bundle branch pacing is achieved at implantation | Baseline (During implantation)
  Defined as a paced (pseudo) right bundle branch block QRS morphology with terminal r/R' in lead V1 and any of the following: i) recording of a LBB potential during intrinsic rhythm (only in patients with normal ventricular activation), ii) transition from non-selective to selective LBBP or non-selective LBBP to LV myocardial capture during decreasing pacing output, iii) abrupt shortening of stimulus to R wave peak time in V6 ECG lead (V6RWPT) ≥10 ms during implantation, iv) V6RWPT < 75ms or < 80ms in patients with preexisting left bundle branch block or v) an interpeak interval (V1RWPT - V6RWPT) ≥ 33ms.
Proportion of patients with left-bundle branch pacing criteria at 24 hours | At 24 hours (before discharge)
  Defined as a paced (pseudo) right bundle branch block QRS morphology with terminal r/R' in lead V1 and any of the following: i) recording of a LBB potential during intrinsic rhythm (only in patients with normal ventricular activation), ii) transition from non-selective to selective LBBP or non-selective LBBP to LV myocardial capture during decreasing pacing output, iii) abrupt shortening of stimulus to R wave peak time in V6 ECG lead (V6RWPT) ≥10 ms during implantation, iv) V6RWPT < 75ms or < 80ms in patients with preexisting left bundle branch block or v) an interpeak interval (V1RWPT - V6RWPT) ≥ 33ms.

SECONDARY OUTCOMES:
Procedural complications | At 24 hours
  Number of patients with major and minor complications related to the procedure (death, perforation, cardiac tamponade, lead dislodgment, loss of capture or need for reintervention)

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro Lorente-Ros, MD, Principal Investigator — Puerta de Hierro University Hospital; Victor Castro-Urda, MD, Study Director — Puerta de Hierro University Hospital
Locations (2):
- Spain (2):
  - Puerta de Hierro University Hospital, Majadahonda, Madrid
  - Fundación Jiménez Díaz University Hospital, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Glikson M, Nielsen JC, Kronborg MB, Michowitz Y, Auricchio A, Barbash IM, Barrabes JA, Boriani G, Braunschweig F, Brignole M, Burri H, Coats AJS, Deharo JC, Delgado V, Diller GP, Israel CW, Keren A, Knops RE, Kotecha D, Leclercq C, Merkely B, Starck C, Thylen I, Tolosana JM; ESC Scientific Document Group. 2021 ESC Guidelines on cardiac pacing and cardiac resynchronization therapy. Eur Heart J. 2021 Sep 14;42(35):3427-3520. doi: 10.1093/eurheartj/ehab364. No abstract available. PMID 34455430
- [Background] Hou X, Qian Z, Wang Y, Qiu Y, Chen X, Jiang H, Jiang Z, Wu H, Zhao Z, Zhou W, Zou J. Feasibility and cardiac synchrony of permanent left bundle branch pacing through the interventricular septum. Europace. 2019 Nov 1;21(11):1694-1702. doi: 10.1093/europace/euz188. PMID 31322651
- [Background] Vijayaraman P, Ponnusamy S, Cano O, Sharma PS, Naperkowski A, Subsposh FA, Moskal P, Bednarek A, Dal Forno AR, Young W, Nanda S, Beer D, Herweg B, Jastrzebski M. Left Bundle Branch Area Pacing for Cardiac Resynchronization Therapy: Results From the International LBBAP Collaborative Study Group. JACC Clin Electrophysiol. 2021 Feb;7(2):135-147. doi: 10.1016/j.jacep.2020.08.015. Epub 2020 Oct 28. PMID 33602393
- [Background] Zhang S, Zhou X, Gold MR. Left Bundle Branch Pacing: JACC Review Topic of the Week. J Am Coll Cardiol. 2019 Dec 17;74(24):3039-3049. doi: 10.1016/j.jacc.2019.10.039. Epub 2019 Dec 9. PMID 31865972
- [Background] Tan JL, Lee JZ, Terrigno V, Saracco B, Saxena S, Krathen J, Hunter K, Cha YM, Russo AM. Outcomes of Left Bundle Branch Area Pacing for Cardiac Resynchronization Therapy: An Updated Systematic Review and Meta-analysis. CJC Open. 2021 Jun 16;3(10):1282-1293. doi: 10.1016/j.cjco.2021.05.019. eCollection 2021 Oct. PMID 34888508
- [Background] De Pooter J, Wauters A, Van Heuverswyn F, Le Polain de Waroux JB. A Guide to Left Bundle Branch Area Pacing Using Stylet-Driven Pacing Leads. Front Cardiovasc Med. 2022 Feb 21;9:844152. doi: 10.3389/fcvm.2022.844152. eCollection 2022. PMID 35265691
- [Background] Braunstein ED, Kagan RD, Olshan DS, Gabriels JK, Thomas G, Ip JE, Markowitz SM, Lerman BB, Liu CF, Cheung JW. Initial experience with stylet-driven versus lumenless lead delivery systems for left bundle branch area pacing. J Cardiovasc Electrophysiol. 2023 Mar;34(3):710-717. doi: 10.1111/jce.15789. Epub 2022 Dec 30. PMID 36571159
- [Background] Shimeno K, Tamura S, Hayashi Y, Abe Y, Naruko T, Fukuda D. Achievement rate and learning curve of left bundle branch capture in left bundle branch area pacing procedure performed to demonstrate output-dependent QRS transition. J Cardiovasc Electrophysiol. 2022 Oct;33(10):2183-2191. doi: 10.1111/jce.15627. Epub 2022 Jul 23. PMID 35842801
- [Background] Huang W, Chen X, Su L, Wu S, Xia X, Vijayaraman P. A beginner's guide to permanent left bundle branch pacing. Heart Rhythm. 2019 Dec;16(12):1791-1796. doi: 10.1016/j.hrthm.2019.06.016. Epub 2019 Jun 22. No abstract available. PMID 31233818